CLINICAL TRIAL: NCT01485406
Title: Safety and Immunogenicity Study of GSK Biologicals' Pneumococcal Vaccine 2830930A When Administered as a Single Dose in Healthy Toddlers Aged 12-23 Months
Brief Title: Safety and Immunogenicity Study of GlaxoSmithKline (GSK) Biologicals' Pneumococcal Vaccine 2830930A Administered in Toddlers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 115373; 2011-002225-22 (EudraCT Number)
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Infections, Streptococcal
Keywords: Haemophilus influenzae; Safety; Pneumococcal vaccine; Streptococcus pneumoniae; Immunogenicity; Toddlers
MeSH Terms: conditions — Streptococcal Infections; Haemophilus Infections | interventions — PHiD-CV vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Pn Group (Experimental): Toddlers 12-23 months of age receiving GSK2830930A vaccine.
  Interventions: Biological: Pneumococcal vaccine GSK2830930A
- Control Group (Active Comparator): Toddlers 12-23 months of age receiving Synflorix.
  Interventions: Biological: Synflorix™

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK2830930A — 1 dose administered intramuscularly
  Arms: Pn Group
Biological: Synflorix™ — 1 dose administered intramuscularly
  Arms: Control Group

SUMMARY:
The purpose of this study is to assess the safety, reactogenicity and immunogenicity of the GSK Biologicals' pneumococcal vaccine 2830930A in toddlers aged 12 to 23 months at study entry.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LARs) can and will comply with the requirements of the protocol.
* A male or female between, and including 12 to 23 months of age at the time of vaccination.
* Written informed consent obtained from the parents/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of at least 36 weeks.
* Previously completed three-dose vaccination course with Synflorix.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/administration of a vaccine containing diphtheria- or tetanus- toxoid or CRM197 and not foreseen by the study protocol during any time of the study period, or of any other vaccines not foreseen by the protocol in the period starting from 30 days before the vaccine dose and ending 30 days after, with the exception of licensed influenza vaccines.

  * The licensed influenza vaccines are always allowed, even if concomitantly administered with the study vaccines but should be documented in the "Concomitant vaccination" of the electronic Case Report Form.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness, including Kawasaki's syndrome.
* History of any neurological disorders or seizures, including conditions such as hypotensive-hyporesponsive episodes, encephalopathy and any convulsions (afebrile and febrile).
* Acute disease and/or fever at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding vaccination or planned administration during study period.
* Any medical condition which might interfere with the assessment of the study objectives in the opinion of the investigator.
* Previous receipt of a booster dose (fourth dose) of Synflorix.
* Anaphylaxis following previous administration of vaccines.

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2011-12-12 (Actual); Primary Completion 2012-03-15 (Actual); Study Completion 2012-03-15 (Actual)

PRIMARY OUTCOMES:
Occurrence of each grade 3 solicited adverse event with relationship to vaccination | Within 7 days (Day 0-Day 6) after vaccination
Occurrence of grade 3 unsolicited adverse events with relationship to vaccination | Within 31 days (Day 0-Day 30) after vaccination
Occurrence of serious adverse events with relationship to vaccination | During the entire study (from Month 0 up to Month 1)

SECONDARY OUTCOMES:
Occurrence of each solicited adverse event | Within 7 days (Day 0-Day 6) after vaccination
Occurrence of each unsolicited adverse event | Within 31 days (Day 0-Day 30) after vaccination
Occurrence of serious adverse event | During the entire study (from Month 0 up to Month 1)
Evaluation of the immune responses to the components of the 2830930A vaccine | One month post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Germany (4):
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Berchtesgaden, Bavaria
  - GSK Investigational Site, Braunatal, Hesse
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20770

REFERENCES:
- [Background] Horn M, Behre U, Traskine M, Dobbelaere K, Borys D. Safety, reactogenicity, and immunogenicity of a 12-valent pneumococcal non-typeable Haemophilus influenzae protein D-conjugate vaccine in healthy toddlers: results from a phase I, randomized trial. Hum Vaccin Immunother. 2021 May 4;17(5):1463-1469. doi: 10.1080/21645515.2020.1810493. Epub 2020 Nov 11. PMID 33175600
- See also: Results for study 115373 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/115373?search=study&b%22b''%22#rs